CLINICAL TRIAL: NCT07161531
Title: Evaluating Test-Retest Reliability of Surface Electromyography (sEMG) in Measuring Fatigue in Adolescents Through Prolonged Activity
Brief Title: Test-retest Reliability of sEMG to Measure Fatigue in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ann Hallemans, Associate Professor, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6979
Record Dates: First submitted 2025-08-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adolescents
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue (Experimental): To induce muscular fatigue, participants will perform a repetitive bodyweight squat until 1) the squat cannot be performed over the full range of motion for 2 consecutive repetitions and 2) physical exertion occurs (10-point Borg scale).
  Interventions: Diagnostic Test: Surface Electromyography

INTERVENTIONS:
Diagnostic Test: Surface Electromyography — The primary lower limb muscles to be monitored include the gluteus medius, rectus femoris, vastus lateralis (quadriceps ), biceps femoris (hamstrings), tibialis anterior, and gastrocnemius medialis (calves). This setup fully utilizes a 16-channel sEMG system by monitoring each muscle group bilaterally to capture comprehensive data on muscle activity and fatigue.

SUMMARY:
This cross-sectional study aims to determine the test-retest reliability of surface electromyography (sEMG) outcomes in detecting levels of fatigue among healthy adolescents engaged in physical activities. It seeks to evaluate the consistency of sEMG parameters across two test sessions and correlate these measurements with both performance metrics and subjective fatigue assessments.

Participants will perform repetitive squatting until volitional exhaustion while their muscular activity is recorded. They will do so on two different test sessions with an interval of one week in between.

ELIGIBILITY:
Inclusion Criteria:

* engage in regular physical activity, such as sports or dance

Exclusion Criteria:

* neuromuscular disorders
* conditions that affect muscle function

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
sEMG median power frequency (MPF) - test | first test session at day 1
  A parameter used to analyze the frequency content of the electrical signals generated by muscle activity. Changes in the MPF can indicate alterations in muscle fiber recruitment and metabolic changes during sustained muscle contractions
sEMG median power frequency - retest | second test session after 1 week
  A parameter used to analyze the frequency content of the electrical signals generated by muscle activity. Changes in the MPF can indicate alterations in muscle fiber recruitment and metabolic changes during sustained muscle contractions
sEMG RMS amplitude - test | first test session at day 1
  A single value that represents the magnitude of the sEMG signal over a specified period of time, higher RMS values indicate greater muscle activation.
sEMG RMS amplitude - retest | second test session after 1 week
  A single value that represents the magnitude of the sEMG signal over a specified period of time, higher RMS values indicate greater muscle activation.

SECONDARY OUTCOMES:
VAS score - test | first test session at day 1
  subjective fatigue score
VAS score - retest | second session after 1 week
  subjective fatigue score

OTHER OUTCOMES:
Age | first test session at day 1
  age in years
Gender | first session
  male/female/other
Height | first test session at day 1
  body height in centimeters
Weight | first test session at day 1
  body weight in kilograms
Leg length | first test session at day 1
  Length measured from trochanter major to the ground in centimeters
Physical Activity | first test session at day 1
  PAQ-A (physical activity questionaire for adolescents): a self-administered, 7-day recall instrument. It was developed to assess general levels of physical activity for high school students in grades 9 to 12 and approximately 14 to 19 years of age.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiteit Antwerpen, Department of Rehabilitation Sciences and Physiotherapy, Research group MOVANT, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mokkink, L.B., de Vet, H., Diemeer, S. et al. Sample size recommendations for studies on reliability and measurement error: an online application based on simulation studies. Health Serv Outcomes Res Method 23, 241-265 (2023)
- [Background] Patikas DA, Williams CA, Ratel S. Exercise-induced fatigue in young people: advances and future perspectives. Eur J Appl Physiol. 2018 May;118(5):899-910. doi: 10.1007/s00421-018-3823-1. Epub 2018 Feb 13. PMID 29441401
- [Background] Lynn SK, Watkins CM, Wong MA, Balfany K, Feeney DF. Validity and Reliability of Surface Electromyography Measurements from a Wearable Athlete Performance System. J Sports Sci Med. 2018 May 14;17(2):205-215. eCollection 2018 Jun. PMID 29769821
- [Background] Cifrek M, Medved V, Tonkovic S, Ostojic S. Surface EMG based muscle fatigue evaluation in biomechanics. Clin Biomech (Bristol). 2009 May;24(4):327-40. doi: 10.1016/j.clinbiomech.2009.01.010. Epub 2009 Mar 13. PMID 19285766

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT07161531/Prot_SAP_000.pdf